CLINICAL TRIAL: NCT01973725
Title: PhaseⅡ Study of Icotinib Hydrochloride in Treating Patients With Recurrent or Metastatic Esophageal Squamous Carcinoma After Failure of Conventional Chemotherapy
Brief Title: Study of Icotinib Hydrochloride in Treating Patients With Recurrent or Metastatic Esophageal Cancer After Failure of Conventional Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-29
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib Hydrochloride (Experimental): Patients will receive Icotinib Hydrochloride at 125mg/times,oral three times daily for 21 days.
  Interventions: Drug: Icotinib Hydrochloride

INTERVENTIONS:
Drug: Icotinib Hydrochloride — Patients will receive Icotinib Hydrochloride at 125mg/times,oral three times daily for 21 days.
  Other Names: Conmana

SUMMARY:
Phase II Study of Icotinib Hydrochloride in Treating Patients With Recurrent or Metastatic Esophageal Squamous Carcinoma After Failure of Conventional Chemotherapy.

DETAILED DESCRIPTION:
Currently,there is no standard second-line therapy for esophageal squamous cell carcinoma.More effective therapy for patients with this disease who developed disease progression after first line therapy is needed.Although Erlotinib is recommended in NCCN Guideline Version 2.2013,there is still insufficient evidence on EGFR-TKI as second-line therapy for esophageal squamous carcinoma.Therefore,further research is necessary.In this phase II study,we evaluate the efficacy and safety of Icotinib Hydrochloride as treatment for patients with recurrent or metastasis esophageal squamous carcinoma after failure of conventional chemotherapy,and analyse the value of biomarkers of these patient to identify who benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form
* Age: 18-75 years old
* Histologically confirmed diagnosis of esophageal squamous cell carcinoma
* Patients have Received and progressed on 1 line of prior Fluoropyrimidine, platinum or taxane based palliative chemotherapy
* Measurable disease in at least 1 diameter by CT scan or MRI as per RECIST 1.1 criteria
* Life expectancy ≥ 3 months
* Karnofsky score ≥70
* Patient has adequate bone marrow and organ function

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 75 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
* Patient has adequate liver function

  * AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis)
  * Serum bilirubin ≤ 2 x ULN
* Creatinine ≤ 1.5 times ULN
* No malabsorption or other gastrointestinal disorders affecting drug absorption.
* No serious complications such as active gastrointestinal hemorrhage, perforation, jaundice, gastrointestinal obstruction, non cancerous fever > 38 ℃.
* Expect good compliance

Exclusion Criteria:

* Patient has received previous treatment with EGFR inhibitors
* Patient is currently receiving Phenytoin, rifampin, barbiturates, C Masi Bing
* Known severe hypersensitivity to Icotinib or any of the excipients of this product
* CNS metastases without radiotherapy and/or surgery
* Patients with treated CNS metastases may participate in this trial,except for those who must receive hormone therapy and those whose prior hormone therapy for CNS metastases is less than 4 weeks
* Evidence of clinically active Interstitial Lung Diseases
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of nonmelanoma skin cancer or cervical carcinoma in situ
* psychiatric illness that would prevent the patient from giving informed consent
* Patient is concurrently using other approved or investigational antineoplastic agent
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disease control rate | for up to 6 months
  Disease control rate of tumor

SECONDARY OUTCOMES:
Overall survival | Time from day 1 to date of death
  From time of diagnosis to death or lost to follow-up
Time to progression | Time from day 1 to date of documented disease progression
  From time of diagnosis to disease progression
Adverse event | Each follow up vist, assessed up to 12 months
  Safety data will be assessed at each study visit using NCI CTCAE version 3.0
EORTC QLQ-C30 and QLQ-OES18 | Time from day 1 to date of death
  Quality of life will be assessed at each study visit using EORTC QLQ-C30 and QLQ-OES18

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuhong, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes